CLINICAL TRIAL: NCT00002944
Title: Chemotherapy for Progressive Low Grade Astrocytoma in Children Less Than Ten Years Old
Brief Title: Combination Chemotherapy in Treating Children With Progressive Brain Tumors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A9952; CCG-A9952 (Other: Children's Cancer Group); POG-A9952 (Other: Pediatric Oncology Group); CCG-9952 (Other: Clinical Trials.gov); CDR0000065394 (Other: Clinical Trials.gov)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-09-09 (Estimated); Status verified 2013-09

CONDITIONS: Brain Tumors; Central Nervous System Tumors
Keywords: recurrent childhood brain stem glioma; recurrent childhood visual pathway glioma; recurrent childhood cerebellar astrocytoma; recurrent childhood cerebral astrocytoma; childhood low-grade cerebellar astrocytoma; childhood low-grade cerebral astrocytoma
MeSH Terms: conditions — Brain Neoplasms; Central Nervous System Neoplasms; Optic Nerve Glioma; Astrocytoma | interventions — Carboplatin; Lomustine; Procarbazine; Thioguanine; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Regimen A (CV Chemotherapy) (Experimental): Induction will consist of 10 weeks of therapy (carboplatin, vincristine sulfate),followed by 2 weeks without chemotherapy. Induction should only be interrupted in the event of grade 3 neurotoxicity, grade 2 renal toxicity, grade 4 hematologic toxicity, or tumor progression. Maintenance-Four Courses (2 cycles/course) commences on Day 84 (week 12) of Induction or when peripheral counts recover with ANC >1,000/$L and platelet count >100,000/$L. Each cycle will consist of 4 weekly doses of carboplatin, three weekly doses of vincristine sulfate (given concomitantly with the first 3 weeks of carboplatin), followed by two weeks of rest for a total of 6 weeks. Maintenance will continue for a total of 8 cycles.
  Interventions: Drug: carboplatin; Drug: vincristine sulfate
- Regimen B (TPCV Chemotherapy) (Experimental): Each cycle of chemotherapy consists of 4 days of oral chemotherapy (Thioguanine, procarbazine hydrochloride, Lomustine and Vincristine sulfate beginning Day 0, followed by vincristine sulfate IV on Days 14 and 28. The cycle is repeated every 6 weeks (42 days). A total of 8 cycles will be given.
  Interventions: Drug: lomustine; Drug: procarbazine hydrochloride; Drug: thioguanine; Drug: vincristine sulfate

INTERVENTIONS:
Drug: carboplatin — Given IV
  Other Names: Paraplatin; NSC-241240
  Arms: Regimen A (CV Chemotherapy)
Drug: lomustine — Given IV
  Other Names: CCNU; NSC-79037
  Arms: Regimen B (TPCV Chemotherapy)
Drug: procarbazine hydrochloride — Given PO
  Other Names: Matulane; NSC-77213
  Arms: Regimen B (TPCV Chemotherapy)
Drug: thioguanine — Given PO
  Other Names: 6-TG; NSC-752
  Arms: Regimen B (TPCV Chemotherapy)
Drug: vincristine sulfate — Given PO and IV
  Other Names: Oncovin; NSC-675574

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: This randomized phase III trial is studying two different combination chemotherapy regimens and comparing how well they work in treating children with low-grade astrocytomas or other residual tumors of the brain.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the event free survival as a result of treatment with carboplatin and vincristine versus thioguanine, procarbazine, lomustine, and vincristine in children with progressive brain tumors.
* Estimate tumor response rates to each regimen of chemotherapy in these patients.
* Determine toxic effects and quality of life of children treated with each regimen of chemotherapy.
* Investigate biological and clinical factors which may predict tumor response and early progression (tumor size, location, pathologic subtype, cytogenetics, and proliferative index by MIB-1 (Ki67)) in these patients.
* Investigate factors contributing to neuropsychological and endocrine status of children with brain tumors treated without irradiation.

OUTLINE: This is a randomized study. Patients are stratified according to site of disease, status at entry, and pathology. Patients are randomized to one of two treatment arms. Patients with neurofibromatosis are nonrandomly assigned to arm II.

* Arm I: Patients receive induction with carboplatin and vincristine for 10 weeks followed by 2 weeks of rest. Induction is followed by 8 courses of maintenance beginning on day 84 of induction or upon hematopoietic recovery. Each course consists of 4 weekly doses of carboplatin and 3 weekly doses of vincristine (given concurrently with the first 3 weeks of carboplatin), followed by 2 weeks of rest.
* Arm II: Patients receive oral thioguanine, procarbazine, and lomustine on days 0-4, followed by vincristine IV on days 14 and 28. Treatment continues every 6 weeks for a maximum of 8 courses.

PROJECTED ACCRUAL: A total of 280-340 patients will be accrued over 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Pathologically confirmed low grade residual astrocytomas or other eligible residual tumors of the brain interpreted as low grade (WHO grades I and II) such as the following:

  * Glial Tumors

    * Astrocytic tumors

      * Low grade astrocytoma (variants: fibrillary, protoplasmic, gemistocytic)
      * Pilocytic astrocytoma
      * Pleomorphic xanthoastrocytomas
      * Subependymal giant cell astrocytoma
      * Infantile desmoplastic astrocytoma
    * Low grade oligodendroglial tumors

      * Low grade oligodendroglioma
    * Low grade mixed gliomas

      * Oligo-astrocytoma
  * Neuronal Tumors

    * Ganglioglioma (excluding tumors with anaplastic astrocytic components)
    * Infantile desmoplastic ganglioglioma
  * Chiasmatic-hypothalamic tumor without histologic confirmation
* All of the following diagnostic tests (radiological or clinical evidence of progression, surgery, or confirmatory MRI) must be carried out within 6 weeks of enrollment into this study
* Progressive disease following surgical excision based on clear radiological or clinical evidence of progression, or an incomplete excision (less than 95% or greater than 1.5 cm2) with necessity to begin treatment because of a risk of neurologic impairment with progression
* Chiasmatic lesions that have contiguous extensions of tumor into other regions of the visual pathways demonstrated on contrast MRI will be eligible for study without histopathological confirmation
* Patients with neurofibromatosis who have radiographic diagnosis of chiasmatic-hypothalamic tumor are eligible for the study, without requiring a biopsy confirmation of tumor histology, but not unless tumor progression is documented radiographically
* No intrinsic brain stem tumors of the pons or isolated optic nerve tumors without definitive involvement of the optic chiasm

PATIENT CHARACTERISTICS:

Age:

* Under 10

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count greater than 1,000/mm^3 (arm II)
* Platelet count greater than 100,000/mm^3 (arm II)

Hepatic:

* Not specified

Renal:

* Creatinine less than 1.5 times upper limit of normal for age OR
* Creatinine clearance or radioisotope GFR greater than 70 mL/min or equivalent GFR as determined by the institutional normal range

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy for the tumor

Endocrine therapy:

* Prior corticosteroid therapy allowed

Radiotherapy:

* No prior radiotherapy for the tumor

Surgery:

* See Disease characteristics

Other:

* Prior diuretic therapy allowed

Max Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 428 (Actual)
Dates: Start 1997-04; Primary Completion 2006-02 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Event Free Survival | Time from study entry until disease progression, death without progression of disease, occurrence of a second malignant neoplasm or last follow-up, whichever comes first, assessed up to 5 years
  Compare the event-free survival as a result of treatment with either CV or TPCV

SECONDARY OUTCOMES:
Survival | 5 years
  Defined as the time to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Joann Ater, MD, Study Chair — M.D. Anderson Cancer Center
Locations (204):
- United States (179):
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Southern California Permanente Medical Group, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Jonathan Jaques Children's Cancer Center at Miller Children's Hospital, Long Beach, California
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Samuel Oschin Comprehensive Cancer Institute at Cedars-Sinai Medical Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Children's Hospital and Research Center Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital at Stanford University Medical Center, Palo Alto, California
  - Sutter Cancer Center, Sacramento, California
  - University of California Davis Cancer Center, Sacramento, California
  - Kaiser Permanente Medical Center - Oakland, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Santa Barbara Cottage Children's Hospital, Santa Barbara, California
  - Kaiser Permanente Medical Center - Santa Clara Kiely Campus, Santa Clara, California
  - Children's Hospital Center for Cancer and Blood Disorders, Aurora, Colorado
  - Carole and Ray Neag Comprehensive Cancer Center at the University of Connecticut Health Center, Farmington, Connecticut
  - Yale Cancer Center, New Haven, Connecticut
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward General Medical Center Cancer Center, Fort Lauderdale, Florida
  - Lee Cancer Care of Lee Memorial Health System, Fort Myers, Florida
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Memorial Cancer Institute at Memorial Regional Hospital, Hollywood, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - Miami Children's Hospital, Miami, Florida
  - Baptist-South Miami Regional Cancer Program, Miami, Florida
  - Florida Hospital Cancer Institute at Florida Hospital Orlando, Orlando, Florida
  - M.D. Anderson Cancer Center at Orlando, Orlando, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Sacred Heart Cancer Center at Sacred Heart Hospital, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - St. Joseph's Cancer Institute at St. Joseph's Hospital, Tampa, Florida
  - Kaplan Cancer Center at St. Mary's Medical Center, West Palm Beach, Florida
  - AFLAC Cancer Center and Blood Disorders Service of Children's Healthcare of Atlanta - Egleston Campus, Atlanta, Georgia
  - AFLAC Cancer Center and Blood Disorders Service of Children's Healthcare of Atlanta - Scottish Rite Campus, Atlanta, Georgia
  - MBCCOP - Medical College of Georgia Cancer Center, Augusta, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - Curtis and Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Mountain States Tumor Institute at St. Luke's Regional Medical Center, Boise, Idaho
  - University of Illinois Cancer Center, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Keyser Family Cancer Center at Advocate Hope Children's Hospital, Oak Lawn, Illinois
  - Advocate Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Swedish-American Regional Cancer Center, Rockford, Illinois
  - Simmons Cooper Cancer Institute, Springfield, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - St. Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - Kosair Children's Hospital, Louisville, Kentucky
  - Tulane Cancer Center Office of Clinical Research, Alexandria, Louisiana
  - Children's Hospital of New Orleans, New Orleans, Louisiana
  - Ochsner Cancer Institute at Ochsner Clinic Foundation, New Orleans, Louisiana
  - CancerCare of Maine at Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program at Barbara Bush Children's Hospital, Scarborough, Maine
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Alvin and Lois Lapidus Cancer Institute at Sinai Hospital, Baltimore, Maryland
  - Dana-Farber/Harvard Cancer Center at Dana-Farber Cancer Institute, Boston, Massachusetts
  - Baystate Regional Cancer Program at D'Amour Center for Cancer Care, Springfield, Massachusetts
  - C.S. Mott Children's Hospital at University of Michigan Medical Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Breslin Cancer Center at Ingham Regional Medical Center, Lansing, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Children's Hospitals and Clinics of Minnesota - St. Paul, Saint Paul, Minnesota
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Keesler Air Force Base Medical Center, Keesler Air Force Base, Mississippi
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Children's Hospital, Omaha, Nebraska
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Hackensack University Medical Center Cancer Center, Hackensack, New Jersey
  - St. Barnabas Medical Center Cancer Center, Livingston, New Jersey
  - Overlook Hospital, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center Hospital, Albany, New York
  - Maimonides Cancer Center at Maimonides Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Don Monti Comprehensive Cancer Center at North Shore University Hospital, Manhasset, New York
  - Schneider Children's Hospital, New Hyde Park, New York
  - Beth Israel Medical Center - Petrie Division, New York, New York
  - NYU Cancer Institute at New York University Medical Center, New York, New York
  - St. Luke's - Roosevelt Hospital Center - St.Luke's Division, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Stony Brook University Cancer Center, Stony Brook, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Dakota Cancer Institute at Dakota Clinic - South University, Fargo, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - Akron Children's Hospital, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's - Dayton, Dayton, Ohio
  - Toledo Hospital, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - Tod Children's Hospital, Youngstown, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Legacy Emanuel Hospital and Health Center and Children's Hospital, Portland, Oregon
  - Knight Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Palmetto Health South Carolina Cancer Center, Columbia, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - East Tennessee Children's Hospital, Knoxville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Sciences Center School of Medicine - Amarillo, Amarillo, Texas
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - Carilion Medical Center for Children at Roanoke Community Hospital, Roanoke, Virginia
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Deaconess Medical Center, Spokane, Washington
  - Providence Cancer Center at Sacred Heart Medical Center, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center - Tacoma, Tacoma, Washington
  - Madigan Army Medical Center - Tacoma, Tacoma, Washington
  - West Virginia University Health Sciences Center - Charleston, Charleston, West Virginia
  - Edwards Comprehensive Cancer Center at Cabell Huntington Hospital, Huntington, West Virginia
  - Mary Babb Randolph Cancer Center at West Virginia University Hospitals, Morgantown, West Virginia
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
- Australia (5):
  - John Hunter Hospital, Newcastle, New South Wales
  - Prince of Wales Private Hospital, Randwick, New South Wales
  - Children's Hospital at Westmead, Westmead, New South Wales
  - Royal Children's Hospital, Brisbane, Queensland
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (16):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Children's & Women's Hospital of British Columbia, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Children's Health and Rehabilitation Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - Children's Hospital of Western Ontario, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Montreal Children's Hospital at McGill University Health Center, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
  - Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan
  - Saskatoon Cancer Centre at the University of Saskatchewan, Saskatoon, Saskatchewan
  - Centre Hospitalier Universitaire de Quebec, Québec
- University Medical Center Groningen, Groningen, Netherlands
- Starship Children's Health, Auckland, New Zealand
- Switzerland (2):
  - Swiss Pediatric Oncology Group Bern, Bern
  - Swiss Pediatric Oncology Group Geneva, Geneva

REFERENCES:
- [Result] Ater JL, Zhou T, Holmes E, Mazewski CM, Booth TN, Freyer DR, Lazarus KH, Packer RJ, Prados M, Sposto R, Vezina G, Wisoff JH, Pollack IF. Randomized study of two chemotherapy regimens for treatment of low-grade glioma in young children: a report from the Children's Oncology Group. J Clin Oncol. 2012 Jul 20;30(21):2641-7. doi: 10.1200/JCO.2011.36.6054. Epub 2012 Jun 4. PMID 22665535